CLINICAL TRIAL: NCT02132507
Title: Multimodal Functional Neuroimaging in Epilepsy Patients
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Other Study IDs: R01EB006433 (NIH); R01EB006433 (NIH)
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Epilepsy
Keywords: epilepsy; fMRI; EEG; ICA
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of the study is to evaluate a new technology for functional neuroimaging using electroencephalography (EEG) and MRI in studying epilepsy.

DETAILED DESCRIPTION:
MRI is a clinical routine test for imaging (creating a picture) of the structure and function of human organs using a giant magnet and other electronic and computing equipment. Functional MRI (fMRI) is an MRI that is done while the subject performs some simple activity or in resting state. It shows the areas of the brain that are activated by performing each of these activities or correlated with spontaneous brain activities (e.g. interictal spikes).

The EEG-fMRI session will be conducted at the University of Minnesota Center for Magnetic Resonance Research. If a subject has any metal implant in his/her body, s/he must not participate in the MRI test. After subjects pass through the routine screening for participation in the MRI test, an EEG cap with 64 electrodes will be put on his/her scalp and electrically conducting gels will be applied to each of these electrodes. One more electrode will be put on his/her back to record electrocardiographic signal. The electrodes location will be recorded by means of a device which can tell the positions of the electrode sensors. The EEG preparation procedure will take around 30-45 minutes. Then a 15-minute EEG will be recorded out side of the scanner. Afterwards, the subject will be asked to lie down in a MRI scanner with the EEG cap on his/her scalp. The electrodes will be connected to a data collection system and electroencephalograms and fMRI will be collected and stored simultaneously onto the computer of the recording system. During the scan, subjects will be asked to close his/her eyes but keep awake. Or subjects may be also asked to perform some simple tasks. For example, subjects may be asked to tap his/her finger regularly or imagine some movements. The EEG-fMRI scan will take around 2 hours. After the recording session, subjects may want to wash his/her hair to clean out the electrically conductive gels. Although the EEG and MRI procedure can be performed as a routine clinical test, in this instance it is being performed for the research and not for his/her clinical care.

Subjects may also be asked to undergo EEG or fMRI recordings separately. In this case, subjects will be asked to perform similar simple tasks as those during EEG-fMRI procedure. The total time involved with either the special EEG session or the MRI (or MRI-EEG) session will be about one to two hours.

Approximately 50 subjects may be involved in this research at the University of Minnesota.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients are diagnosed with medically intractable epilepsy;
* 2. patients have frequent interictal spikes on clinical EEG monitorings;
* 3. patients without large morphological abnormalities

Exclusion Criteria:

* Patients with skull bony defects, intracerebral mass lesions, major brain malformations, large cystic regions will be excluded.
* Any indwelling metal objects or implantable devices such as pace makers, cochlear implants, or implanted intracranial electrodes.
* Patients with claustrophobia.
* Patients with more than 2 grand mal seizures per month.
* Patients will not be excluded on the basis of location of seizure onset zone, type or number of medications, or cognitive status (assuming the minimum criteria has been met), or race.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are seen at the epilepsy center of School of medicine, University of Minnesota
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2011-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Localization of epileptogenic foci | 12/31/2014
  Finding of epileptogenic foci in patients with focal epilepsy

CONTACTS AND LOCATIONS:
Overall Officials: Bin He, PhD, Principal Investigator — Distinguished McKnight University Professor of Biomedical Engineering Medtronic-Bakken Chair for Engineering in Medicine Director, Institute for Engineering in Medicine Director, Center for Neuroengineering
Locations (1):
- Biomedical Engineering Department, Minneapolis, Minnesota, United States